CLINICAL TRIAL: NCT02828163
Title: Comparative Study Between Intralesional Autologous Platelet Rich Plasma and Intralesional Triamcinolone Acetonide in the Oral Erosions of Pemphigus Vulgaris Patients
Brief Title: Comparison Between Injections of Steroids and Autologous Platelet Rich Plasma in the Oral Erosions of Pemphigus Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwah Adly Saleh, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP # steroids in pemphigus
Record Dates: First submitted 2016-06-27; First posted 2016-07-11 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Oral Pemphigus Vulgaris
MeSH Terms: interventions — Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous Platelet rich plasma (Experimental): Autologous platelet-rich plasma (PRP) is autologous plasma that has platelet concentration above the baseline. 1 millilitre of autologous platelet-rich plasma will be injected in one side of the oral mucosa of pemphigus vulgaris patients every 2 weeks for 3 months.
  Interventions: Other: Autologous Platelet rich plasma
- Triamcinolone acetonide (Active Comparator): Triamcinolone acetonide is an effective treatment for oral erosions of pemphigus vulgaris patients. 10mg/ml of Triamcinolone acetonide will be injected in one side of the oral mucosa of pemphigus vulgaris patients every 2 weeks for 3 months.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Other: Autologous Platelet rich plasma — Intralesional injection of 1 milliliter of autologous Platelet rich plasma in the oral erosions every 2 weeks for 3 months.
  Other Names: autologous PRP
  Arms: Autologous Platelet rich plasma
Drug: Triamcinolone Acetonide — 10mg/ml of Triamcinolone acetonide will be injected in one side of the oral mucosa of pemphigus vulgaris patients every 2 weeks for 3 months.
  Other Names: Kenacort
  Arms: Triamcinolone acetonide

SUMMARY:
Comparing the effect of injecting autologous platelet rich plasma and triamcinolone acetonide in the erosions of buccal mucosa of pemphigus vulgaris patients.

DETAILED DESCRIPTION:
Ten (Pemphigus vulgaris (PV) patients will be enrolled in this study. The clinical disease score of the patients will be assessed using the pemphigus disease area index (PDAI). Three milliliters of blood will be withdrawn from each patient. The blood will be centrifuged and the platelet rich plasma (PRP) will be extracted. Patients will receive autologous PRP injections for one side of buccal mucosa and triamcinolone acetonide 10mg/ml at the other buccal mucosa at biweekly intervals for 3 months. The degree of pain and clinical improvement of each buccal mucosa will be assessed by an investigator who does not know the nature of injection in each buccal mucosa. Therefore the investigation doing the injection will not be blind but the other investigator assessing the results will be blind also the patients will be blind.

ELIGIBILITY:
Inclusion Criteria:

* Pemphigus vulgaris patients having bilateral erosions in the buccal mucosa.

Exclusion Criteria:

* Pemphigus vulgaris patients who do not have oral erosions.
* Pemphigus vulgaris patients who have received intralesional steroid injection in their buccal mucosa.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Improvement of the size of oral erosions. | 3 months
  These observations will be performed at start and end of treatment period by evaluating patients's photos by two blinded observers. The clinically measured score of improvement will be recorded by both observers. Score of improvement is defined as 0-25% clinical improvement of ulcers = poor response to treatment, 26-50% clinical improvement of ulcers = average response, 51-75% clinical improvement of ulcers = good response, >75% excellent response
Improvement of the depth of oral erosions. | 3 months
Improvement of the degree of erythema of oral erosions. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed HM EL-Komy, M.D, Study Chair — Dermatology Department Cairo University
Locations (1):
- Faculty of Medicine Cairo University Dermatology Department, Cairo, Please Select, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] EL-Komy MH, Hassan AS, Abdel Raheem HM, Doss SS, EL-Kaliouby M, Saleh NA, Saleh MA. Platelet-rich plasma for resistant oral erosions of pemphigus vulgaris: A pilot study. Wound Repair Regen. 2015 Nov-Dec;23(6):953-5. doi: 10.1111/wrr.12363. Epub 2015 Nov 4. PMID 26340377
- [Background] Saleh MA. Pemphigus in the Arab world. J Dermatol. 2015 Jan;42(1):27-30. doi: 10.1111/1346-8138.12676. PMID 25558949
- [Background] Mignogna MD, Fortuna G, Leuci S, Adamo D, Dell'Aversana Orabona G, Ruoppo E. Adjuvant triamcinolone acetonide injections in oro-pharyngeal pemphigus vulgaris. J Eur Acad Dermatol Venereol. 2010 Oct;24(10):1157-65. doi: 10.1111/j.1468-3083.2010.03610.x. PMID 20236381